CLINICAL TRIAL: NCT06526091
Title: Cerebral Oxygen Saturation Monitoring During Optimum Cord Management in Preterm (COSMIC Pilot Study)
Brief Title: Cerebral Oxygen Saturation Monitoring During Optimum Cord Management in Preterm Infants
Acronym: COSMIC
Status: Recruiting | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22QC7933
Record Dates: First submitted 2022-08-26; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Pre-Term
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants: Preterm infants born at less than 34 completed weeks gestation
  Interventions: Other: Cerebral NIRS monitoring at delivery

INTERVENTIONS:
Other: Cerebral NIRS monitoring at delivery — Application of cerebral NIRS monitoring immediately after delivery and during optimum cord management

SUMMARY:
This study will assess the feasibilty measuring cerebral oxygen saturations using a Near Infrared Spectroscopy (NIRS) monitor immediately after delivery of preterm infants. The investigators aim to evaluate the effects of optimum cord management on cerebral oxygenation in this cohort

DETAILED DESCRIPTION:
Optimal cord management is defined by delaying clamping of the umbilical cord for 1 minute after delivery and is recommend in all neonates, regardless of gestational age. Transfusion of blood from placenta to baby in this minute enables smooth cardiovascular transition and stable cerebral perfusion. Preterm infants are at increased risk of haemodynamic instability and brain injury if the cord is clamped too early. It remains unclear what the optimum time is to clamp the cord in preterm infants, and it is likely different for each baby. Current monitoring of heart rate and peripheral oxygen saturations does not correlate well with oxygen delivery to the brain. Near infrared spectroscopy (NIRS) is a non-invasive method of measuring regional cerebral oxygenation saturations. NIRS may be a helpful monitoring tool to guide optimum timing of cord clamping in preterm infants.

This study aims to assess the feasibility of using the INVOS 5100 NIRS monitor immediately after delivery in preterm infants born before 34 weeks gestational age. The investigators aim to assess if they can generate meaningful data on brain oxygen levels in the first few minutes of life. The secondary objectives are to use this data to describe the changes in heart rate, peripheral oxygen and cerebral oxygen saturations during placental transfusion and cord clamping.

The investigators will use the INVOS device to measure cerebral oxygenation immediately after delivery, during placental transfusion and cord clamping. We will assess the feasibility of the INVOS device for this purpose. We will use the INVOS data and routinely collected data at delivery to evaluate the effect of optimum cord management on cerebral perfusion, heart rate and peripheral oxygen saturations.

ELIGIBILITY:
Inclusion Criteria:

* All babies eligible for optimum cord management born before 34 completed weeks gestational age
* Parental consent

Exclusion Criteria:

* Multiple pregnancies
* Infants for whom resuscitation at birth is not appropriate
* Antenatal or immediate postnatal diagnosis of severe congenital anomaly
* Infants with complex congenital cardiac disease

Ages: 1 Minute to 24 Hours | Sex: All
Age Groups: Child
Study Population: Preterm infants born at less than 34 completed weeks gestational age at Queen Charlotte and Chelsea Hospital (London) undergoing optimum cord management during birth
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of regional cerebral saturation (rSO2 in %) monitoring using NIRS during optimum cord | 2 years
  Feasibility of regional cerebral saturation (rSO2 in %) monitoring using NIRS during optimum cord management in preterm infants

SECONDARY OUTCOMES:
Arterial saturation (SaO2 in %) monitoring | 2 years
  Evaluating the effect of optimum cord management on SaO2
Oxygenation (FiO2 in %) during stabilisation | 2 years
  Evaluating the effect of preterm stabilisation including optimum cord management on FiO2 (%)

CONTACTS AND LOCATIONS:
Overall Officials: Jayanta Banerjee, MD (Res), Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No